CLINICAL TRIAL: NCT03079375
Title: The Impact of Pharmaceutical Medication Review, Medication Interview Before Discharge and Follow-up: A Randomized Controlled Trial
Brief Title: The Pharmacist Follows You and Your Medication From Hospital to Your Daily Life and Investigate What This Means to You
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lene V. Ravn-Nielsen (Other)
Collaborators: The Hospitals Pharmacies' and Amgros' Research Development Foundation (Unknown); University of Southern Denmark (Other); Two public Regional foundations (Unknown); The Actavis Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Lene V. Ravn-Nielsen, Clinical pharmacist, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: Cross-sectorial medicine
Record Dates: First submitted 2017-03-01; First posted 2017-03-14 (Actual); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Cross-Sectional Study
Keywords: cross sectional; medication review; readmissions; follow-up

STUDY DESIGN:
Intervention Model Description: The combination of pharmacist interventions are compared with medication review alone in comparison to non-intervention (a control group).
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The study is double blinded. The pharmacist do not know, whether the patient is randomized to the basic or to the extended intervention before they conduct the medication review. That is why the patients in the intervention group are randomized two times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- usual care (No Intervention): no pharmaceutical intervention.
- basic intervention (Sham Comparator): Medication review
  Interventions: Other: basic intervention
- extended intervention (Sham Comparator): medication review, medication interview before discharge and follow-up with patient, GP and if relevant pharmacy and nursing home.
  Interventions: Other: extended intervention

INTERVENTIONS:
Other: basic intervention — medication review
  Arms: basic intervention
Other: extended intervention — medication review, medication interview before discharge and follow-up
  Arms: extended intervention

SUMMARY:
Background

It is well known that the transfer of a patient from hospital to the general practitioner is related with mistakes in the medication of the patient. A report from 2006 measure the number of drug related admissions in Denmark to be 69.000 to 162.000 per year. To reduce these mistakes, more and better communication between the health professionals are suggested. Furthermore medication reviews made by pharmacist seems to reduce the number of drug related readmissions and other drug related issues, which can lead to an economic cost reduction.

Objective

The aim of this study is to investigate the impact of medication review and better communication between the health professionals after discharge of a patient from hospital to the general practitioner. The effect is measured as reducing the number of readmissions and number of visits at the emergency department 30 days and six month after inclusion of the patient.

Method

This study was estimated to include 1500 participants. The patients were randomized to one of three groups; usual care, basic intervention or extended intervention. The usual care received the normal care following the Danish standard procedure. The basic intervention had a medication review by a clinical pharmacist during admission.

The extended interventions group was similar to the basic intervention group plus follow-up with the patient, the general practitioner and if relevant the nursing home and pharmacy one week and six month after discharge by interview with the clinical pharmacist.

DETAILED DESCRIPTION:
The aim of this study is to determine if a multifaceted pharmacist intervention based on medication review, medication interview and follow up with patient, general practitioner and pharmacy can reduce the number of readmissions and death and or if the time to next admission can be postponed. The combination of the full pharmacist intervention is compared with medication review alone in comparison to non-intervention.

Pharmacist intervention:

Usual care group: the patients received no intervention by the clinical pharmacist.

Basic intervention group: A structured, patient centered medication review (MR) was conducted by the clinical pharmacist. The following was considered during MR: Were there untreated diagnoses, has the goal of treatment been reached, was the treatment compliant with current national guidelines regarding dose, choice of drug and time of treatment. Focus was at certain drugs most commonly implicated in causing admission. Furthermore, all drugs on the medication list were assessed according to the following: Indication for treatment, drug dose, considering i.e. kidney insufficiency, age, etc., adverse drug events, therapeutic duplication, dosage time and interval, drug formulation and strength, interactions, contraindications, precautions and specific patient characteristics.

Advice on drug selection, dosages, monitoring needs and possibly side effects were given to the physician in charge of the patient, and written in the electronic patient journal (EPJ).

Extended intervention group: MR was conducted according to the same terms and conditions as for the basic intervention group. Upon discharge medication reconciliation was conducted. The pharmacist provided a motivational interview (MI)-based patient interview including a comprehensive summary of changes in the drug therapy during the hospitalization.

Post discharge any drug related problem not dealt with during hospitalization was mailed or faxed to the general practitioner (GP). When needed, the GP, care giver and primary care pharmacy were contacted by phone (approximately five working days after discharge).

Follow-up interview by phone was performed twice. The first was conducted one week post discharge and the second six months after discharge. When needed additional follow-ups could be made. The follow-up interviews had an motivational interview approach.

All interventions were conducted according to a defined standard operating procedure and all interventions were performed by qualified clinical pharmacists from the involved sites. In order to minimize the risk of cultural differences and variations in routine's the regions in between, all data pharmacists were trained prior to entering the study.

Data was analysed after the intention-to-treat method. Data was analyzed after a proportional hazard cox regression with the randomization group as the only variable.

ELIGIBILITY:
Inclusion Criteria:

* Usual medicine of five drugs or above
* Speak and understand Danish
* Admitted via the Acute Medicine Admission Ward
* Are able to give informed consent

Exclusion Criteria:

* Patients included in a similar study
* Declared terminal
* Suicidal
* In custody
* Isolated at the hospital
* Im- and/or expressive aphasia
* Severe dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1499 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2015-04-24 (Actual); Study Completion 2015-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lene V. Ravn-Nielsen, M.Sc.Pharm, Study Director — Hospital Pharmacy of Funen

IPD SHARING:
Plan to Share IPD: Yes
Only during data analysis between clinical pharmacists. Personal identification number is converted to an anonymous identification number.

REFERENCES:
- [Derived] Ravn-Nielsen LV, Duckert ML, Lund ML, Henriksen JP, Nielsen ML, Eriksen CS, Buck TC, Pottegard A, Hansen MR, Hallas J. Effect of an In-Hospital Multifaceted Clinical Pharmacist Intervention on the Risk of Readmission: A Randomized Clinical Trial. JAMA Intern Med. 2018 Mar 1;178(3):375-382. doi: 10.1001/jamainternmed.2017.8274. PMID 29379953

RESULTS

PARTICIPANT FLOW:
Groups:
- Extended Intervention: medication review, medication interview before discharge and follow-up with patient, general practitioner and if relevant pharmacy and nursing home.
  extended intervention: medication review, medication interview before discharge and follow-up
Period: Overall Study
Arm/Group | Usual Care | Basic Intervention | Extended Intervention
Started | 503 | 499 | 497
Completed | 498 | 493 | 476
Not Completed | 5 | 6 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Basic Intervention | Extended Intervention | Total
Number analyzed (Participants) | 498 | 493 | 476 | 1467
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 121 | 141 | 130 | 392
  >=65 years | 377 | 352 | 346 | 1075
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73 [65 to 80] | 72 [63 to 80] | 71 [63 to 79] | 72 [63 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 278 | 248 | 262 | 788
  Male | 220 | 245 | 214 | 679
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Readmissions
Description: number of patients who have been readmitted
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Basic Intervention | Extended Intervention
Number analyzed (Participants) | 498 | 493 | 476
Participants | 111 | 98 | 68

2. Primary Outcome: Admissions
Description: number of patients who have been admitted
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Basic Intervention | Extended Intervention
Number analyzed (Participants) | 498 | 493 | 476
Participants | 243 | 233 | 189

3. Primary Outcome: Emergency Department Visits
Description: number of patients who have emergency department visits
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Basic Intervention | Extended Intervention
Number analyzed (Participants) | 498 | 493 | 476
Participants | 21 | 19 | 15

4. Primary Outcome: Composite Endpoint, Admissions or Emergency Department Visits
Description: number of patients who experience primary composite endpoint, admissions or emergency department visits within 6 month
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Basic Intervention | Extended Intervention
Number analyzed (Participants) | 498 | 493 | 476
Participants | 243 | 233 | 193

5. Secondary Outcome: Drug-related Admissions
Description: number of patients who have drug related admissions
Time Frame: 180 days after the inclusion date
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Basic Intervention | Extended Intervention
Number analyzed (Participants) | 498 | 493 | 476
Participants | 96 | 95 | 75

6. Secondary Outcome: Drug-related Readmissions
Description: number of patients who have drug related readmissions
Time Frame: 30 days after the inclusion date
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Basic Intervention | Extended Intervention
Number analyzed (Participants) | 498 | 493 | 476
Participants | 38 | 34 | 24

7. Secondary Outcome: Percentage of Medication Changes Accepted by GPs
Description: Acceptance rate in primary care (general practitioner). Medication review data were not collected from the Usual care Group and were collected only for the Basic and Extended Groups.
Time Frame: up to 180 days
Population: Medication review data were not collected from the Usual care Group and were collected only for the Basic and Extended Groups. No interventions were sent to the general practitioner for the Usual care and the Basic intervention Groups.
Measure: Number; unit: percentage of medication changes
Arm/Group | Extended Intervention
Number analyzed (Participants) | 476
percentage of medication changes | 66

8. Secondary Outcome: Medication Review Changes Accepted by Physicians (in Hospital)
Description: Medication review data were not collected from the Usual care Group and were collected only for the Basic and Extended Groups.
Time Frame: 1 month
Population: Medication review data were not collected from the Usual care Group and were collected only for the Basic and Extended Groups. The acceptance rate is only analyzed for of the basic intervention and the extended intervention in total.
Measure: Number; unit: percentage of medication changes
Arm/Group | Basic Intervention | Extended Intervention
Number analyzed (Participants) | 493 | 476
percentage of medication changes | 61 | 61

9. Secondary Outcome: Mortality
Description: number of patient who died within 6 month after inclusion
Time Frame: 180 days after the inclusion date
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Basic Intervention | Extended Intervention
Number analyzed (Participants) | 498 | 493 | 476
Participants | 50 | 42 | 54

10. Secondary Outcome: Drug Related Mortality
Description: number of patients who have drug related death
Time Frame: 180 days after the inclusion date
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Basic Intervention | Extended Intervention
Number analyzed (Participants) | 498 | 493 | 476
Participants | 6 | 3 | 5

ADVERSE EVENTS:
Time Frame: 6 months
Description: The adverse event data was not collected because the Danish medicines agency found that the study did not require registration of adverse events according to Danish law.
Arm/Group | Usual Care | Basic Intervention | Extended Intervention
All-Cause Mortality (participants affected / at risk) | 50/498 | 42/493 | 54/476
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes